CLINICAL TRIAL: NCT02644382
Title: Improving Surgical Decision-making in Young Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shoshana M. Rosenberg, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 15-288; 1K01HS023680-01A1 (AHRQ)
Record Dates: First submitted 2015-12-20; First posted 2015-12-31 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; decision making; surgery; qualitative
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Decision Support Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Key Informant interviews: 20 in-person or phone qualitative interviews with patients.
  Interventions: Other: qualitative data collection
- Focus Groups: four qualitative focus groups of 6-10 women each.
  Interventions: Other: qualitative data collection
- Physician Interviews: physician qualitative interviews over the telephone.
  Interventions: Other: qualitative data collection
- Usual care cohort (pilot): 50 women who will be surveyed before and after their surgical consult
  Interventions: Other: survey
- Decision aid cohort (pilot): 50 women who will be surveyed before and after their surgical consult and will also be sent a web-based decision aid
  Interventions: Other: survey; Other: decision aid

INTERVENTIONS:
Other: qualitative data collection — qualitative data collection
  Groups: Focus Groups; Key Informant interviews; Physician Interviews
Other: survey — survey pre and post-surgical consult
  Groups: Decision aid cohort (pilot); Usual care cohort (pilot)
Other: decision aid — web-based decision aid post-surgical consult
  Groups: Decision aid cohort (pilot)

SUMMARY:
The overall goal of this study is to qualitatively assess the surgical decision-making process from both the patient and physician perspective

1. Conduct short in-person interviews with young women prior to surgery
2. Conduct focus groups with breast cancer survivors about their surgical decision and experience
3. Interview surgical oncologists, plastic surgeons, medical and radiation oncologists about their experiences and how they communicate with breast cancer patients about local therapy decisions
4. To survey women about surgical decision-making prior to and after their consult in conjunction with pilot testing of a web-based decision aid to support high quality surgical decision-making in newly diagnosed young women with breast cancer.

DETAILED DESCRIPTION:
Breast cancer in young women: Breast cancer is the most common cancer diagnosed in women younger than age 40 in the United States, with approximately 14,000 new cases each year. Young women face unique psychosocial challenges, most notably fertility, sexuality, and image concerns and are at a life stage where education, career, and family are important priorities. Concern about these issues may contribute to the greater psychosocial distress seen in younger women at both diagnosis and in follow-up compared with older women. Importantly, these concerns may also influence treatment decisions including receipt of chemotherapy, adherence to endocrine therapy, and surgical decisions. Thus, attending to the unique issues of young women may enhance not only quality of care and quality of life (QOL) but also potentially disease outcomes.

Surgical management of breast cancer: Standard loco-regional management of breast cancer entails partial mastectomy (i.e., breast conserving surgery) followed by radiation or mastectomy with or without radiation. The decision depends on a number of factors including extent of disease, family history, BRCA mutation status, and personal preference. In recent years, an increasing number of women have elected to undergo contralateral prophylactic mastectomy (CPM) in conjunction with surgery of the affected breast (usually choosing bilateral mastectomy), despite a lack of clear evidence for survival benefit from this procedure in the vast majority of women. In weighing the benefits and risks of CPM, one must consider the absolute risk reduction of a new primary breast cancer (usually relatively modest in the average risk survivor), the long and short-term risks of this additional surgery including potential complications (bilateral mastectomy is associated with a greater risk of surgical complications) and the impact on QOL. At the same time, one must consider the competing risk of systemic recurrence of a woman's initial breast cancer. Young women, in particular, have the greatest risk of systemic recurrence and death from their original cancer, lowering the likelihood of benefit of CPM in preventing a new primary breast cancer. However, while CPM rates have increased among all breast cancer patients, increased rates of CPM are particularly pronounced among the youngest women with breast cancer, with several studies identifying young age at diagnosis as one of the strongest determinants of CPM.Physicians and researchers have been observing and discussing this trend for a number of years and yet little has been done to intervene.

The goal of the proposed research is to better understand and improve the surgical decision process in young women with breast cancer. Using qualitative research methods, we will comprehensively assess patient experiences - both patients who have had CPM and patients who did not - as well as physician perspectives regarding this decision. Based on these findings, the investigators will determine how to best improve the quality of the process, e.g., by correcting misperceptions, setting realistic expectations regarding the impact of surgery (including reconstruction) on QOL, improving communication with health care providers, and better management of anxiety surrounding diagnosis. This qualitative research is designed to build on prior quantitative analyses, by gaining an in depth perspective through focus groups and interviews, about certain issues identified as impacting the surgical decision process, including anxiety, fear of recurrence, and patient-physician communication.

Collectively, results from the qualitative assessment will inform a future phase of this research involving the design and subsequent development of a decision aid to help women make informed decisions about their breast cancer surgery.

The goal of this second phase of the research is to survey women about surgical decision-making prior to and after their consult in conjunction with pilot testing of a web-based decision aid to support high quality surgical decision-making in newly diagnosed young women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients for key informant interviews-

1. Newly diagnosed women with Stage 0-3 breast cancer
2. Between the ages of 18 and 40 who are seen at DFCI and have not yet had their primary breast cancer surgery.

Patients for focus groups:

1. diagnosis of Stage 0-3 breast cancer at age 40 and younger
2. currently between the ages of 18-43
3. English-speaking
4. 1-3 years from diagnosis
5. Had breast cancer surgery
6. no evidence of recurrent or metastatic disease.

Providers:

Must care for women who have breast cancer. Can be surgeons, surgical oncologists, medical and/or radiation oncologists

Patients for Surgical Decision Making Pilot

1. Women with newly-diagnosed, unilateral Stage 0-3 breast cancer
2. Between the ages of 18 and 40
3. Who are seen by a surgeon at DFCI/BWH or Faulkner Hospital
4. English speaking
5. Have not yet had their primary breast cancer surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young Women with a history of breast cancer and providers who care for them.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Thematic summary from the data gathered from the use of a moderator guide (series of probing questions) that inquires about the experiences surrounding the surgical decision-making process from both the patient and physician perspective | 1 year
  The goal of the proposed research is to better understand and improve the surgical decision process in young women with breast cancer. Using qualitative research methods, we will comprehensively assess patient experiences - both patients who have had CPM and patients who did not - as well as physician perspectives regarding this decision.
Breast cancer knowledge | 2 weeks
  Knowledge will be assessed using selected questions from the Breast Cancer Surgery Decision Quality Instrument (BCS-DQI), an instrument designed to evaluate the quality of breast cancer treatment decisions as well as additional true/false questions related to side effects of radiation.
Decisional conflict | 2 weeks
  Decisional conflict will be measured with the SURE scale. The SURE scale is composed of four items from the Decisional Conflict Scale that measure patients' uncertainty about which treatment choice and factors contributing to uncertainty.
Anxiety | 2 weeks
  Anxiety will be assessed using the PROMIS Emotional Distress - Anxiety - Short Form.
Treatment goals and preferences | 2 weeks
  have been adapted from the BCS-DQI. We will ask women to mark on a scale (not important - very important) the importance of several reasons in relation to their decision about surgery as well as concerns (not all concerned-very concerned) about local therapy.
Perception of decision process | 2 weeks
  Perception of the decision process will be assessed with an adapted version of the Control Preferences Scale.

SECONDARY OUTCOMES:
Usability of decision aid (DA) | 2 weeks-1 month
  Assessment of what patients did and did not like about the DA, ways they think the DA can be improved, and how they felt the DA affected communication with their physician.

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Rosenberg, ScD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg SM, Greaney ML, Patenaude AF, Sepucha KR, Meyer ME, Partridge AH. "I don't want to take chances.": A qualitative exploration of surgical decision making in young breast cancer survivors. Psychooncology. 2018 Jun;27(6):1524-1529. doi: 10.1002/pon.4683. Epub 2018 Apr 6. PMID 29476578
- [Background] Rosenberg SM, Greaney ML, Patenaude AF, Partridge AH. Factors Affecting Surgical Decisions in Newly Diagnosed Young Women with Early-Stage Breast Cancer. J Adolesc Young Adult Oncol. 2019 Aug;8(4):463-468. doi: 10.1089/jayao.2019.0002. Epub 2019 Apr 3. PMID 30942651